CLINICAL TRIAL: NCT06314399
Title: Predictive Factors Associated with Bile Culture Positivity and PhenotypiCal AntIbiogram Resistance Patterns in Patients Taken to LaparOscopic Cholecystectomy (BACILO): a Protocol for a Prediction Model Study
Brief Title: Predictive Factors Associated to Bile Cultures and Antibiogram Resistance in Patients with Laparoscopic Cholecystectomy
Acronym: BACILO
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Mayor Méderi (Other)
Collaborators: Universidad del Rosario (Other)
Responsible Party: Principal Investigator, Camilo Ramirez Giraldo, Principal Investigator - General Surgeon, Hospital Universitario Mayor Méderi
Other Study IDs: 2023-18; DVO005 2555-CV1837 (Other: Universidad del Rosario Research Ethics Committee)
Record Dates: First submitted 2024-03-08; First posted 2024-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-03

CONDITIONS: Biliary Infection; Antibiotic Resistant Strain
Keywords: biliary infection; bactibilia; antibiotic resistance; laparoscopic cholecystectomy
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3-5cm of bile will be extracted from the surgical specimen (gallbladder), during laparoscopic cholecystectomy to be taken for bacterial cultures and phenotypical antibiogram resistance pattern if it is positive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Bile culture and phenotypic antibiogram resistance test — Extraction of 3-5ml of bile from surgical specimen (gallbladder) to be taken for bacterial culture testing and phenotypical antibiogram resistance if positive

SUMMARY:
The BACILO study was designed with the objective of having robust data on local epidemiological bacterial colonisation information on bile cultures with patients taken to laparoscopic cholecystectomy in our institution to find which predictive factors are associated with culture positivity and antibiotic resistance patterns. Secondary endpoints include evaluating demographical, clinical and surgical variables and establishing comparison between both positive and negative bile cultures and between antibiotic sensitive and resistant microorganism strain isolations.

DETAILED DESCRIPTION:
BACILO is single-centre, observational, analytical, prospective study with a prognostic prediction model with the objective of identifying predictive factors associated with microbial and antibiotic resistance patterns in bile cultures of patients taken to laparoscopic cholecystectomy in our institution. Primary outcomes are bile culture positivity and phenotypical resistance antibiogram patterns while secondary outcomes include demographic, clinical and surgical characteristics and surgical outcomes. The main objective is to determine predictive factors using a prediction model, variables included are: Age, diabetes mellitus, C-reactive protein test, choledocholithiasis/ERCP, cholecystitis and severity of cholecystitis according to the 2018 Tokyo guidelines.This in the nature of describing the relationship between bile culture positivity and phenotypical antibiogram resistance patterns in our institution, and establish thus better treatment strategies based on higher quality local evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients included must be over 18 years of age and be taken to laparoscopic cholecystectomy between March 2024 and February 2026 in any institution of the Méderi hospital network (Hospital Universitario Mayor and Hospital Universitario Barrios Unidos), have signed the written informed consent to be included in the study and have both bile culture and antibiogram.

Exclusion Criteria:

* - Patients that will be taken to laparoscopic cholecystectomy with another concomitant surgical procedure (including but not exclusive to gastrectomy, pancreatoduodenectomy, oesophagectomy, splenectomy, abdominal wall reconstruction, colectomy, amongst others) with the exception of umbilical herniorrhaphy.
* Patients without a postoperative control appointment.
* Patients with an untreated HIV diagnosis.
* Patients with diagnosis of a malignant gallbladder or biliary tract disease documented preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are over 18 years that have an indication for laparoscopic cholecystectomy in our institution without any of the exclusion criteria, which had bile cultures taken from the surgical specimen (gallbladder) during the surgery and attended the postoperative15 day follow-up appointment after hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Bile culture positivity | Perioperatively, during the procedure and immediately after the intervention
  Bile culture is tested positive for at least one (1) microorganism
Phenotypical antibiogram resistance | Perioperatively, during the procedure and immediately after the intervention
  If bile culture is positive, evaluation for possible antibiotic resistance vs sensitivity

SECONDARY OUTCOMES:
Microbial characteristics | Immediately after the intervention
  To describe the microbial characteristics of the bile cultures and their phenotypical antibiogram resistance
Bile culture and antibiotic resistance relationship | Immediately after the intervention
  Explore the relationship between positive bile cultures and phenotypical antibiogram resistance with surgical outcomes
Demographical and clinical characteristics | Pre-intervention
  To describe and compare the demographic and clinical characteristics of the study population.
Surgical characteristics and outcomes | During the 15 day postoperative follow-up appointment
  To describe and compare the surgical characteristics and outcomes of the study population
Determination of predictive factors (age, diabetes mellitus, choledocholithiasis / ERCP, C-reactive protein, cholecystitis and Tokyo guidelines severity of cholecystitis) | Through study completion, around 1 year and a half
  To determine demographic and clinical predictive factors for positive bile cultures and phenotypical antibiogram resistance.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Hospital Universitario Mayor-Méderi, Bogota, Cundinamarca
  - Hospital Universitario Méderi Barrios Unidos, Bogota, Cundinamarca

IPD SHARING:
Plan to Share IPD: Yes
Data obtained and input into the database is anonymous, without any individual or identifying characteristics will be stored in a dataset from the Centro de Recursos para el Aprendizaje y la Investigación, property of and administered by the Universidad del Rosario as a plan of data management. Moreover, the different codes used in the analysis will be stored in this dataset.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It is in our plans once we obtain a register number from Clinical Trials in order to publish the protocol, statistical analysis plan and clinical study report in a scientific journal so it will be available to all people interested.
Access Criteria: It is in our plans to be published in a scientific journal available to all people interested.

REFERENCES:
- [Background] Dyrhovden R, Ovrebo KK, Nordahl MV, Nygaard RM, Ulvestad E, Kommedal O. Bacteria and fungi in acute cholecystitis. A prospective study comparing next generation sequencing to culture. J Infect. 2020 Jan;80(1):16-23. doi: 10.1016/j.jinf.2019.09.015. Epub 2019 Oct 2. PMID 31586461
- [Background] Pisano M, Allievi N, Gurusamy K, Borzellino G, Cimbanassi S, Boerna D, Coccolini F, Tufo A, Di Martino M, Leung J, Sartelli M, Ceresoli M, Maier RV, Poiasina E, De Angelis N, Magnone S, Fugazzola P, Paolillo C, Coimbra R, Di Saverio S, De Simone B, Weber DG, Sakakushev BE, Lucianetti A, Kirkpatrick AW, Fraga GP, Wani I, Biffl WL, Chiara O, Abu-Zidan F, Moore EE, Leppaniemi A, Kluger Y, Catena F, Ansaloni L. 2020 World Society of Emergency Surgery updated guidelines for the diagnosis and treatment of acute calculus cholecystitis. World J Emerg Surg. 2020 Nov 5;15(1):61. doi: 10.1186/s13017-020-00336-x. PMID 33153472
- [Background] Galili O, Eldar S Jr, Matter I, Madi H, Brodsky A, Galis I, Eldar S Sr. The effect of bactibilia on the course and outcome of laparoscopic cholecystectomy. Eur J Clin Microbiol Infect Dis. 2008 Sep;27(9):797-803. doi: 10.1007/s10096-008-0504-8. Epub 2008 Mar 28. PMID 18369670
- [Background] Yoon JH, Paik KY, Chung HY, Oh JS. Clinical implication of bactibilia in moderate to severe acute cholecystitis undergone cholecystostomy following cholecystectomy. Sci Rep. 2021 Jun 4;11(1):11864. doi: 10.1038/s41598-021-91261-9. PMID 34088947
- [Background] van der Linden YT, Bosscha K, Prins HA, Lips DJ. Single-port laparoscopic cholecystectomy vs standard laparoscopic cholecystectomy: A non-randomized, age-matched single center trial. World J Gastrointest Surg. 2015 Aug 27;7(8):145-51. doi: 10.4240/wjgs.v7.i8.145. PMID 26328034
- [Background] Gomi H, Solomkin JS, Schlossberg D, Okamoto K, Takada T, Strasberg SM, Ukai T, Endo I, Iwashita Y, Hibi T, Pitt HA, Matsunaga N, Takamori Y, Umezawa A, Asai K, Suzuki K, Han HS, Hwang TL, Mori Y, Yoon YS, Huang WS, Belli G, Dervenis C, Yokoe M, Kiriyama S, Itoi T, Jagannath P, Garden OJ, Miura F, de Santibanes E, Shikata S, Noguchi Y, Wada K, Honda G, Supe AN, Yoshida M, Mayumi T, Gouma DJ, Deziel DJ, Liau KH, Chen MF, Liu KH, Su CH, Chan ACW, Yoon DS, Choi IS, Jonas E, Chen XP, Fan ST, Ker CG, Gimenez ME, Kitano S, Inomata M, Mukai S, Higuchi R, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: antimicrobial therapy for acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):3-16. doi: 10.1002/jhbp.518. Epub 2018 Jan 9. PMID 29090866
- [Background] Wu ZY, Wu XS, Yao WY, Wang XF, Quan ZW, Gong W. [Pathogens' distribution and changes of antimicrobial resistance in the bile of acute biliary tract infection patients]. Zhonghua Wai Ke Za Zhi. 2021 Jan 1;59(1):24-31. doi: 10.3760/cma.j.cn112139-20200717-00559. Chinese. PMID 33412630
- [Background] Manrai M, Jha AA, Singh Shergill SP, Thareja S, Sood AK, Shukla R, Jain R, Dhiman P, Gaurab. Microbiology of bile in extrahepatic biliary obstruction: A tropical experience. Indian J Med Microbiol. 2021 Jan;39(1):54-58. doi: 10.1016/j.ijmmb.2020.10.002. Epub 2020 Dec 4. PMID 33610257
- [Background] Lee JM, Kang JS, Choi YJ, Byun Y, Jin SH, Yoon KC, Lee HW, Jang JY, Lim CS. Suggested use of empirical antibiotics in acute cholecystitis based on bile microbiology and antibiotic susceptibility. HPB (Oxford). 2023 May;25(5):568-576. doi: 10.1016/j.hpb.2023.01.017. Epub 2023 Feb 3. PMID 36804057
- [Background] Kaplan U, Handler C, Chazan B, Weiner N, Hatoum OA, Yanovskay A, Kopelman D. The Bacteriology of Acute Cholecystitis: Comparison of Bile Cultures and Clinical Outcomes in Diabetic and Non-Diabetic Patients. World J Surg. 2021 Aug;45(8):2426-2431. doi: 10.1007/s00268-021-06107-2. Epub 2021 Apr 15. PMID 33860354
- [Background] Shafagh S, Rohani SH, Hajian A. Biliary infection; distribution of species and antibiogram study. Ann Med Surg (Lond). 2021 Sep 7;70:102822. doi: 10.1016/j.amsu.2021.102822. eCollection 2021 Oct. PMID 34540214
- [Background] Jang DK, Kim J, Park WB, Yi SY, Lee JK, Yoon WJ. Increasing burden of biliary tract infection caused by extended-spectrum beta-lactamase-producing organisms in Korea: A nationwide population-based study. J Gastroenterol Hepatol. 2020 Jan;35(1):56-64. doi: 10.1111/jgh.14809. Epub 2019 Aug 13. PMID 31359494
- [Derived] Ramirez-Giraldo C, Rodriguez Barbosa C, Isaza-Restrepo A, Avendano-Morales V, Rojas-Lopez S, Van-Londono I. Predictive factors associated with Bile culture positivity And phenotypiCal antIbiogram resistance patterns in patients taken to LaparOscopic cholecystectomy (BACILO): protocol for a prospective observational cohort study and development of a prognostic prediction model. BMJ Open. 2024 Nov 1;14(10):e086655. doi: 10.1136/bmjopen-2024-086655. PMID 39486833